CLINICAL TRIAL: NCT07103746
Title: Study of Ublituximab in Early, Active, Autoantibody-Positive, IMMune-MedIated NecroTizing Myopathy (AIM01)
Brief Title: Ublituximab in Autoantibody Positive Immune Mediated Necrotizing Myopathy
Acronym: SUMMIT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (Other); TG Therapeutics (Unknown); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DAIT AIM01
Record Dates: First submitted 2025-07-21; First posted 2025-08-05 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Autoimmune Disorders
Keywords: Ublituximab; Active Autoantibody Positive Immune-Mediated Necrotizing Myopathy (IMNM); Idiopathic inflammatory myopathies (IIM)
MeSH Terms: conditions — Autoimmune Diseases; Myositis | interventions — ublituximab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Initial Ublituximab Active Group (Experimental): Receives 150 mg Ublituximab at Day 0 and 450 mg Ublituximab at Week 2, followed by 450 mgs of Ublituximab at Weeks 24 and 48.
  At Week 26, will receive a Placebo dose of 450 mg to maintain the blind.
  Interventions: Drug: Ublituximab; Drug: Placebo for Ublituximab
- Initial Placebo of ublituximab Group (Experimental): Receives 150 mg Placebo at Day 0 and 450 mg Placebo at Week 2. Receives 150 mg Ublituximab at Week 24 followed by 450 mg Ublituximab at Weeks 26 and 48.
  Interventions: Drug: Ublituximab; Drug: Placebo for Ublituximab

INTERVENTIONS:
Drug: Ublituximab — Initial dose includes 150 mg dose followed by 450 mg two weeks later; maintenance dose is 450 mg
  Other Names: BRIUMVI(TM)
Drug: Placebo for Ublituximab — 0.9% sodium chloride injection

SUMMARY:
This is a multi-center, Phase 2 trial of ublituximab as first-line combination therapy in early, active autoantibody positive immune-mediated necrotizing myopathy.

The primary objective is to estimate the effect of ublituximab as first add-on combination therapy at 24 weeks compared to placebo in treating early, active autoantibody positive immune-mediated necrotizing myopathy using the validated 2016 American College of Rheumatology/ European League Against Rheumatism (ACR/EULAR) Myositis Response Criteria, as measured by the Total Improvement Score (TIS)

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be able to understand and provide informed consent.
2. Age 18 years or older at disease onset.
3. Definite or probable IIM per the 2017 EULAR/ACR classification criteria.
4. Diagnosis of IMNM, meeting the 2016 ENMC classification criteria and having either of the following antibodies:

   1. Anti-SRP
   2. Anti-HMGCR
5. Early disease as defined as onset of objective muscle weakness assessed by a physician and/or CK elevation attributed to IMNM within 1 year of the time of informed consent.
6. Muscle weakness as assessed by an MMT-8 score < 142 of 150 and CK > 1.5x ULN along with abnormality in at least 1 of the following 4 CSMs at screening:

   1. PhGA ≥ 2 cm
   2. PtGA ≥ 2 cm
   3. Extramuscular global assessment ≥ 2 cm
   4. HAQ-DI ≥ 0.25
7. Only one background immunosuppressant treatment for IMNM. Permitted background therapy includes:

   a. Exactly one of the following with medication type stable for at least 12 weeks prior to randomization, and medication dose stable for at least 4 weeks prior to randomization: methotrexate up to 25 mg/weekly, mycophenolate mofetil up to 3000 mg/daily, mycophenolic acid up to 2160 mg/daily, azathioprine up to 2.5 mg/kg daily, tacrolimus up to 0.2 mg/kg daily, or cyclosporine up to 5 mg/kg daily.
8. Current therapy consisting of glucocorticoid ≤ 20 mg/day of prednisone. The dose must be stable for at least 4 weeks prior to randomization. Participants who stopped treatment with glucocorticoids are eligible if the last dose of the glucocorticoids was at least 4 weeks before the time of informed consent.
9. Female participants of childbearing potential and male participants with a partner of childbearing potential must agree to consistently and correctly use FDA approved highly effective methods of birth control, as shown in Appendix 1: Acceptable Contraception Methods for Females of Reproductive Potential, for the entire duration of the study and 6 months after last study drug infusion. Female participants of reproductive potential must have a negative pregnancy test at screening and at baseline.

Exclusion Criteria:

1. End-stage myositis with end-organ involvement that poses additional risk to the participant or confounds the assessment of the participant in the study. Conditions include but are not limited to advanced symptomatic interstitial lung disease (e.g., Forced Vital Capacity (FVC) <60% and/or requiring oxygen therapy) or severe dysphagia.
2. Irreversible muscle involvement and/or severe atrophy that will pose additional risk to the participant or confound the assessment of the participant in the study. This includes Muscle Damage VAS ≥ 3 cm at screening, documented history of severe atrophy of multiple muscle groups (based on MRI), and/or wheelchair bound.
3. Uncontrolled interstitial lung disease or any other uncontrolled IIM manifestation that in the opinion of the investigator would be likely to require treatment with prohibited medication during the study.
4. Diagnosis of other inflammatory or noninflammatory myopathies, including antibody-negative IMNM, inclusion body myositis, overlap myositis, metabolic myopathies, muscular dystrophies or family history of muscular dystrophy, drug induced, cancer-associated myositis, or endocrine-based myositis (except statin induced anti-HMGCR associated IMNM).
5. Severe liver disease, such as signs of ascites or hepatic encephalopathy.
6. History of malignancy (excluding non-melanoma skin cancer) unless cured by adequate treatment, with no evidence of recurrence for ≥ 5 years before the first administration of the study drug.
7. Recent or ongoing bacterial, viral, or fungal infection requiring systemic treatment within 14 days of the time of informed consent.
8. Current suppressive therapy for any chronic infections including herpes simplex virus (HSV).
9. Infection with Mycobacterium tuberculosis (TB) as defined by any of the following:

   1. Positive interferon gamma release assay (IGRA) performed at screening or within 12 weeks prior to the time of informed consent.
   2. Indeterminate IGRAs must be repeated (with same or other IGRA per local policy) and shown to be negative. Alternatively, if the assay remains indeterminant, a participant must have a negative purified protein derivative (PPD) skin test. Finally, if the participant has had the Bacille Calmette-Guerin (BCG) vaccine or has some other condition complicating the interpretation of TB testing, consultation with infectious disease specialist must be obtained before randomization.
10. Medical history or serologic evidence at screening of chronic infections, including:

    a. Human immunodeficiency virus (HIV) infection b. Hepatitis B virus (HBV) as indicated by surface antigen or hepatitis B core antibody positivity c. Hepatitis C virus (HCV) as indicated by anti-hepatitis C antibody positivity. If a participant is Hepatitis C antibody positive, they will be eligible to participate in the study if they have a negative viral load at Screening.
11. Known hypersensitivity reaction to ublituximab.
12. Received a live or live-attenuated vaccine < 4 weeks before the time of informed consent. Received any other type of vaccine < 2 weeks before the time of informed consent.
13. Any of the following laboratory tests at screening:

    a. Hemoglobin < 10 g/dL b. Absolute white blood cell count < 3,000 cells/mm3 c. Platelet count < 100,000 cells/mm3 d. Absolute neutrophils < 1,500 cell/mm3 e. Peripheral B-cell < 5/µL f. IgG < 690 mg/dL g. Estimated GFR < 50 mL/min/1.73 m2
14. Treatment with any immunosuppressive or immunomodulatory agent, such as cyclophosphamide, biologics, and Janus kinase (JAK) inhibitors, except those listed in the inclusion criteria 7 within 12 weeks prior to randomization.
15. Prior receipt of B-cell depleting agents such as rituximab, ocrelizumab, ofatumumab, or belimumab at any time.
16. Treatment of IMNM with IVIG or subcutaneous immunoglobulin (SCIG) within 12 weeks of randomization, or prior receipt of more than one cycle of IVIG at any time.
17. Participant has current or history (within 12 months of screening) of alcohol, drug, or medication abuse.
18. Participant is pregnant or lactating or intends to become pregnant during the study.
19. Use of any investigational drug within 24 weeks of the time of informed consent.
20. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements, or that may impact the quality or interpretation of the data obtained from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is the Total Improvement Score (TIS) at Week 24 reflecting the change from baseline | At 24 weeks
  TIS is a composite endpoint based on improvement in the 6 Disease Activity Core Set Measure (CSM) scores and ranges from 0 to 100 (2016 American College of Rheumatology [ACR] Myositis Response Criteria/European League Against Rheumatism [EULAR]). A higher score indicates more improvement.

SECONDARY OUTCOMES:
Change in mean Total Improvement Score (TIS) value | From baseline to weeks 48, 60, and 72
  Defined as achieving the Total Improvement Score (TIS)
Proportion of participants achieving minimal improvement response (TIS >= 20 points) | From baseline to weeks 24, 48, 60 and 72
  Defined as achieving The Total Improvement Score (TIS) > =20 points (minimum improvement) and >= 40 points (moderate improvement)
Proportion of participants achieving moderate improvement response (TIS >= 40 points) | From baseline to weeks 24, 48, 60 and 72
  Defined as achieving The Total Improvement Score (TIS) > =20 points (minimum improvement) and >= 40 points (moderate improvement)
Time to achieving minimal improvement response (TIS >= 20 points) | From baseline to week 24
  Defined as achieving The Total Improvement Score (TIS) > =20 points (minimum improvement) and >= 40 points (moderate improvement)
Time to achieving moderate improvement response (TIS >= 40 points) | From baseline to week 24
  Defined as achieving The Total Improvement Score (TIS) > =20 points (minimum improvement) and >= 40 points (moderate improvement)
Proportion of participants meeting the definition of worsening | At week 24, 48, 60, and 72
Change from baseline in muscle endurance | At week 24, 48, 60, and 72
  As measured by Functional index-3 scores (FI-3)
Change from baseline in Creatine Kinase (CK) value | At week 24, 48, 60 and 72
Change from baseline in proximal Manual Muscle Testing (MMT) | At week 24, 48, 60, and 72
  As measured by testing the following muscles: trapezius, deltoid, biceps, iliopsoas, gluteus maximum, gluteus medius, quadriceps
Incidence of treatment-emergent adverse events (TEAEs) | From baseline to week 24
Incidence of serious adverse events (SAEs) | From baseline to week 24
Incidence of adverse events (AEs) leading to treatment discontinuation | From baseline to week 24
Change from baseline in the serum autoantibody titers | At week 24, 48, 60 and 72
Change from baseline in peripheral B-cells | At week 24, 48, 60 and 72
Change from baseline in cytokine levels | At week 24, 48, 60 and 72

CONTACTS AND LOCATIONS:
Overall Officials: Julie Paik, M.D., M.H.S., Study Chair — Johns Hopkins Hospital: Division of Rheumatology
Locations (2):
- United States (2):
  - Johns Hopkins Hospital: Division of Rheumatology, Baltimore, Maryland
  - University of Texas - Houston, Houston, Texas

REFERENCES:
- See also: Autoimmunity Centers of Excellence (ACE) — https://www.autoimmunitycenters.org/
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — http://www.niaid.nih.gov/about/dait